CLINICAL TRIAL: NCT00489177
Title: Optimal Programming to Improve Mechanical Indices, Symptoms and Exercise in Cardiac Resynchronization Therapy.
Acronym: OPTIMISE-CRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Dr. Derek Exner, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 73-1726
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy; response; Defibrillators
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): QuickOpt
  Interventions: Device: A
- B (Placebo Comparator): Usual care
  Interventions: Device: B

INTERVENTIONS:
Device: A — QuickOpt intra-cardiac electrogram optimization
  Arms: A
Device: B — Single optimization in initial month post-implant
  Arms: B

SUMMARY:
This international study is assessing if repeat adjustment of the timing between the three leads in a cardiac resynchronization therapy (CRT) defibrillator will increase the likelihood of benefit (symptoms and heart function) compared to usual device programming. The hypothesis is that QuickOpt facilitated serial optimization of sensed atrioventricular (sAV), paced atrioventricular (pAV), and inter-ventricular (VV) timing in the initial 9 months following successful CRT will increase the rate of clinical response and structural remodeling at 12 months compared to usual care.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is primarily designed to synchronize the mechanical activity of the heart. While CRT is beneficial in average, a sizable proportion of patients do not clearly benefit from (respond to) CRT. Whether routinely optimizing the timing between the atria and ventricles (AV timing) and the timing between the left and right ventricles (VV timing) will significantly increase the likelihood of patients benefiting from (responding to) CRT is unknown.

The combination of simple and reliable measures of functional capacity (specific activity score [SAS] and 6-minute walk distance) with echocardiographic measures of left ventricular (LV) volume and ejection fraction (EF) is a practical way of defining response to CRT.

Based on surveys, most patients receiving CRT devices do not have formal optimization of AV and VV timing. This is largely because the usefulness of this is questionable and significant resources are required to perform detailed echo measurements.

A method for estimating optimal sensed AV (sAV), paced AV (pAV), and VV timing using intra-cardiac electrograms (I-EGM) has been developed (QuickOptTM) and offers a quick, simple and inexpensive means to optimize both CRT timing. However, the utility of QuickOptTM optimization is unproven.

Primary hypothesis. QuickOpt facilitated serial optimization of sAV, pAV, and VV timing in the initial 9 months following successful CRT will increase the rate of clinical response and structural remodeling at 12 months compared to usual care. Clinical response will be defined as a reduction in SAS of > 1 class or a 25% or larger improvement in 6 minute hall walk distance at 12 months versus baseline. Structural remodeling will be defined as a 15% or greater reduction in left LV end systolic volume or ≥ 5% absolute improvement in echo-derived LV EF at 12 months versus baseline.

Methods. Initially a sub-study of FREEDOM (NCT00418314). Now an independent trial. Double-blind randomized comparison of serial QuickOpt optimization of sAV, pAV, and VV timing (QuickOpt) versus usual care (Usual) in patients with highly symptomatic heart failure undergoing CRT implantation. Stratification by etiology of LV dysfunction will be undertaken. Serial optimization of sAV, pAV, and VV timing will be performed in the QuickOptTM group immediately post-randomization, and at 3, 6, and 9 months post-randomization. Final outcome will be assessed at 12 months post-randomization.

Statistical aspects. 450 patients (225 / group) will provide 85% power to detect a 15% absolute improvement in the rate of response to CRT with QuickOptTM versus usual care. The proportion of responders will be compared using a Mantel-Haenszel stratified analysis adjusted for lead position (anterior versus non-anterior) and using an intention-to-treat analysis.

Overview. Up to 50 sites in Canada, Europe, Asia and the United States will enroll patients over 36 months. Countries presently enrolling patients include: Canada, the United States, Switzerland, Italy, Belgium, Denmark, Austria, France, Spain, the United Kingdom, the Netherlands, China, Hong Kong and Japan.

ELIGIBILITY:
Inclusion Criteria:

1. CRT-D indications and be implanted with an SJM CRT-D device with VV timing and a compatible lead system.
2. Able to complete a 6-minute hall walk with the only limiting factor to be fatigue or shortness of breath.
3. Geographically stable and willing to comply with follow-up.
4. Adequate echocardiographic images to measure LV end systolic volume.

Exclusion Criteria:

1. Epicardial ventricular lead system.
2. Ability to walk ≥ 450 meters in 6 minutes
3. Limited intrinsic atrial activity (≤ 40 bpm).
4. Persistent or permanent AF.
5. 2° or 3° heart block.
6. Life expectancy is less than 1 year.
7. Patient is pregnant.
8. Receiving IV inotropic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2007-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical benefit (reduction in SAS of at least 1 class or a 25% or larger improvement in 6 minute hall walk distance) plus structural remodeling (15% or greater reduction in left LV end systolic volume or ≥ 5% absolute improvement in echo-derived LV EF) | 12 months

SECONDARY OUTCOMES:
Rate of late (12-month) versus early (3 month) response to CRT | 3 and 12 months
Changes in BNP | 3 and 12 months
Inter-/intra-ventricular dysynchrony | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada